CLINICAL TRIAL: NCT03986463
Title: CIrculating Tumour DNA in Lung Cancer (CITaDeL): Optimizing Sensitivity and Clinical Utility
Acronym: CITaDeL
Status: Completed | Type: Observational
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Other Study IDs: CITaDeL
Record Dates: First submitted 2019-04-30; First posted 2019-06-14 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2020-08

CONDITIONS: Lung Neoplasms; Lung Cancer; Neoplasm of Lung; Non Small Cell Lung Cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Circulating tumour DNA (ctDNA) will be isolated from blood samples and stored for potential future testing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cohort 1: 1. Stage III NSCLC as per the American Joint Committee on Cancer 8th edition (AJCC 8th ed.)
  2. Appropriate to undergo concurrent chemotherapy and radiation
  3. Planned radiation dose must be between 54 and 66 Gy
  4. Chemotherapy regimen must include a platinum agent plus one of the following doublet agents: etoposide, pemetrexed, paclitaxel, vinorelbine, docetaxel, gemcitabine or vincristine
  5. Day 1 platinum dose must be ≥ carboplatin 1.6 AUC or cisplatin 30 mg/m2
  6. No prior system chemotherapy (induction) for their stage III NSCLC, any adjuvant chemotherapy given for resected disease must have been at least 100 days prior to enrollment
  Interventions: Other: Circulating tumour DNA (ctDNA)
- Cohort 2: 1. Stage IV NSCLC or stage III NSCLC, as per the AJCC 8th ed.
  2. Planning to start systemic cytotoxic chemotherapy, without concurrent radiation
  3. Previous treatment with tyrosine kinase inhibitors or immunotherapy (PD-1, PD-L1, CTLA4 directed antibodies) is allowed as long as no cytotoxic chemotherapy was given concurrently
  4. Previous palliative radiation is permitted, but must have been completed at least at least 21 days prior to the initiation of treatment
  5. Chemotherapy regimen must include a platinum agent plus one of the following doublet agents: etoposide, pemetrexed, paclitaxel, vinorelbine, docetaxel, gemcitabine or vincristine
  6. Day 1 platinum dose must be ≥ carboplatin 1.6 AUC or cisplatin 30 mg/m2
  7. If cytotoxic chemotherapy was previously given for adjuvant or stage III NSCLC it must have been at least 100 days prior to enrollment
  Interventions: Other: Circulating tumour DNA (ctDNA)
- Cohort 3: 1. Patients with advanced NSCLC set to undergo palliative radiation to the primary or regional or distant metastatic lesion(s), including intracranial lesions
  2. Radiation dose scheduling must be 2.5 to 4.0 Gy on days 1 through 3 for extracranial treatment, ideally 40 Gy in 15 fractions, 20 Gy in 5 fractions, or 30 Gy in 10 fractions.
  3. Radiation dose for brain lesions must be 6 to 9 Gy per dose, ideally 30 to 35 Gy in 5 daily fractions or 27 Gy in 3 fractions on alternating days
  4. No plans for concurrent chemotherapy to be given
  5. Five patients in cohort 3 will receive radiation to the primary tumor and five patients will receive radiation to brain lesions
  Interventions: Other: Circulating tumour DNA (ctDNA)

INTERVENTIONS:
Other: Circulating tumour DNA (ctDNA) — Circulating tumour DNA (ctDNA) will be isolated from blood samples

SUMMARY:
This is a prospective observation study in patients with non-small cell lung cancer (NSCLC) starting either cytotoxic chemotherapy or radiation therapy. It will assess changes in circulating tumor DNA (ctDNA) in the days following the initiation of treatment, as well as longitudinal monitoring, to assess the dynamics and value of ctDNA in stage III-IV NSCLC.

DETAILED DESCRIPTION:
The study consists of three cohorts of patients initiating a new treatment for their NSCLC. The cohorts of (1) patients starting concurrent chemotherapy and radiation for stage III NSCLC (2) patients with advanced NSCLC starting cytotoxic chemotherapy (with or without pembrolizumab) (3) patients with advanced NSCLC starting palliative radiation therapy. This study aims to study the changes in ctDNA levels following a new treatment in lung cancer patients and to explore if the diagnostic utility of ctDNA testing is improved immediately following treatment when tumour cells are actively dying. It will also examine the changes in ctDNA levels and mutational analysis longitudinally.

ELIGIBILITY:
Inclusion Criteria:

* Histologically diagnosed NSCLC
* Age 18 or older
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-3
* Patients must be able to provide informed consent
* Patients must meet the criteria above AND fulfill the criteria below for entry into one of the 3 cohorts

Cohort 1

1. Stage III NSCLC as per the American Joint Committee on Cancer 8th edition (AJCC 8th ed.)
2. Appropriate to undergo concurrent chemotherapy and radiation
3. Planned radiation dose must be between 54 and 66 Gy
4. Chemotherapy regimen must include a platinum agent plus one of the following doublet agents: etoposide, pemetrexed, paclitaxel, vinorelbine, docetaxel, gemcitabine or vincristine
5. Day 1 platinum dose must be ≥ carboplatin 1.6 AUC or cisplatin 30 mg/m2
6. No prior system chemotherapy (induction) for their stage III NSCLC, any adjuvant chemotherapy given for resected disease must have been at least 100 days prior to enrollment

Cohort 2

1. Stage IV NSCLC or stage III NSCLC, as per the AJCC 8th ed.
2. Planning to start systemic cytotoxic chemotherapy, without concurrent radiation
3. Previous treatment with tyrosine kinase inhibitors or immunotherapy (PD-1, PD-L1, CTLA4 directed antibodies) is allowed as long as no cytotoxic chemotherapy was given concurrently
4. Previous palliative radiation is permitted, but must have been completed at least at least 21 days prior to the initiation of treatment
5. Chemotherapy regimen must include a platinum agent plus one of the following doublet agents: etoposide, pemetrexed, paclitaxel, vinorelbine, docetaxel, gemcitabine or vincristine
6. Day 1 platinum dose must be ≥ carboplatin 1.6 AUC or cisplatin 30 mg/m2
7. If cytotoxic chemotherapy was previously given for adjuvant or stage III NSCLC it must have been at least 100 days prior to enrollment

Cohort 3

1. Patients with advanced NSCLC set to undergo palliative radiation to the primary or regional or distant metastatic lesion(s), including intracranial lesions
2. Radiation dose scheduling must be 2.5 to 4.0 Gy on days 1 through 3 for extracranial treatment, ideally 40 Gy in 15 fractions, 20 Gy in 5 fractions, or 30 Gy in 10 fractions.
3. Radiation dose for brain lesions must be 6 to 9 Gy per dose, ideally 30 to 35 Gy in 5 daily fractions or 27 Gy in 3 fractions on alternating days
4. No plans for concurrent chemotherapy to be given
5. Five patients in cohort 3 will receive radiation to the primary tumor and five patients will receive radiation to brain lesions

Exclusion Criteria:

* Any other malignancy in the last five years other than adequately treated non-melanoma skin cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving treatment at the London Regional Cancer Program in London, Ontario, Canada.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
To measure the change in quantitative ctDNA levels following the initiation of cytotoxic chemotherapy or radiation | Cohort 1 and 2: Baseline (pre-treatment) to end of cycle 1 (each cycle is 21 days) of chemotherapy. Cohort 3: Baseline (pre-treatment) to end of radiotherapy (up to 3 weeks)
  Post-treatment ctDNA levels will be reported as the mean percent increase with standard deviation at maximum compared to baseline (pre-treatment) ctDNA levels.
To identify the timepoint after the initiation of treatment at which the quantified level of ctDNA peaks | Cohort 1 and 2: Baseline (pre-treatment) to end of cycle 1 (each cycle is 21 days) of chemotherapy. Cohort 3: Baseline (pre-treatment) to end of radiotherapy (up to 3 weeks)
  This will be reported as the mean time to maximal ctDNA level with standard deviation from the initiation of treatment
To detect genetic alterations at the time point of maximal ctDNA that were not present in baseline testing | Cohort 1 and 2: Baseline (pre-treatment) to end of cycle 1 (each cycle is 21 days) of chemotherapy. Cohort 3: Baseline (pre-treatment) to end of radiotherapy (up to 3 weeks)
  Will be reported as gene names, with allelic frequencies, found in post-treatment samples that were not present in samples collected at baseline.

SECONDARY OUTCOMES:
To identify the proportion of patients that do not have genetic alterations present in baseline samples but have genetic alterations detected at the timepoint of maximal quantified ctDNA | Cohort 1 and 2: Baseline (pre-treatment) to end of cycle 1 (each cycle is 21 days) of chemotherapy. Cohort 3: Baseline (pre-treatment) to end of radiotherapy (up to 3 weeks)
  This will be reported as frequency counts and proportions.
To determine the percentage of stage III patients with clinically relevant (targetable or prognostic), at any stage of lung cancer, ctDNA genetic alterations. | Cohort 1 and 2: Baseline (pre-treatment) to end of cycle 1 (each cycle is 21 days) of chemotherapy. Cohort 3: Baseline (pre-treatment) to end of radiotherapy (up to 3 weeks)
  Will be reported as frequency counts and proportions.

CONTACTS AND LOCATIONS:
Locations (1):
- London Regional Cancer Program, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Breadner DA, Vincent MD, Correa R, Black M, Warner A, Sanatani M, Bhat V, Morris C, Jones G, Allan A, Palma DA, Raphael J. Exploitation of treatment induced tumor lysis to enhance the sensitivity of ctDNA analysis: A first-in-human pilot study. Lung Cancer. 2022 Mar;165:145-151. doi: 10.1016/j.lungcan.2022.01.013. Epub 2022 Jan 29. PMID 35124411